CLINICAL TRIAL: NCT01280942
Title: Early Warning System for Clinical Deterioration on General Hospital Wards.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 10-0514; 7322-01 (Other Grant/Funding Number: BJH Foundation/ICTS)
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Escalation of Care; Cardiopulmonary Arrest; Respiratory Arrest; Severe Sepsis; Septic Shock
Keywords: clinical deterioration; detection algorithms; automated warning systems
MeSH Terms: conditions — Heart Arrest; Apnea; Sepsis; Shock, Septic; Clinical Deterioration

STUDY DESIGN:
Intervention Model Description: Random allocation of study wards to intervention and control, with washout period and crossover of assignment.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients admitted to 4 GHWs designated as controls. Nurses will not be notified when patients on these GHWs satisfy the EWS algorithm. They will also not wear the wireless sensor devices.
- Nurse notification of EWS alert (Experimental): Patients admitted to 4 GHWs designated as intervention wards at BJH. Nurses will be notified when patients on these wards satisfy the EWS algorithm. Some patients will be asked to wear the wireless remote sensors.
  Interventions: Behavioral: EWS Nursing Alerts; Device: Wireless Remote Sensor

INTERVENTIONS:
Behavioral: EWS Nursing Alerts — An automated algorithm (EWS) will identify patients at potential risk of clinical deterioration. When a patient satisfies the algorithm, a nurse on the patient's ward will be notified. S/he will assess the patient and institute any interventions that are clinically required.
  Arms: Nurse notification of EWS alert
Device: Wireless Remote Sensor — A subset of patients will be consented to wear a wireless sensor device which will monitor heart rate and level of oxygen in the blood.
  Arms: Nurse notification of EWS alert

SUMMARY:
The goal is to develop a two-tiered monitoring system to improve the care of patients at risk for clinical deterioration on general hospital wards (GHWs) at Barnes-Jewish Hospital (BJH). The investigators hypothesize that the use of an automated early warning system (EWS) that identifies patients at risk of clinical deterioration, with notification of nurses on the GHWs when patients are identified, will reduce the risk of ICU transfer or death within 24 hrs of an alert. As a substudy, the investigators will pilot the use of a wireless pulse oximeter to establish feasibility and to develop algorithms for a real-time event detection system (RDS) in these high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 and above, hospitalized in GHWs at Barnes Jewish Hospital.

Exclusion Criteria:

* Minors, patients younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20031 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Bailey, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Result] Bailey TC, Chen Y, Mao Y, Lu C, Hackmann G, Micek ST, Heard KM, Faulkner KM, Kollef MH. A trial of a real-time alert for clinical deterioration in patients hospitalized on general medical wards. J Hosp Med. 2013 May;8(5):236-42. doi: 10.1002/jhm.2009. Epub 2013 Feb 25. PMID 23440923

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Nurse Notification of EWS Alert
Started | 10120 | 9911
Completed | 10120 | 9911
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Nurse Notification of EWS Alert | Total
Number analyzed (Participants) | 10120 | 9911 | 20031
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [44 to 69] | 57 [44 to 70] | 57 [44 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5355 | 5308 | 10663
  Male | 4765 | 4603 | 9368
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4864 | 4790 | 9654
  White | 5062 | 4934 | 9996
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 194 | 187 | 381
Region of Enrollment [Number; unit: participants]
  United States | 10120 | 9911 | 20031

OUTCOME MEASURES:

1. Primary Outcome: Transfer to ICU or Unexpected Death Within 24 Hrs of Identification by the EWS Algorithm
Description: The proportion of patients transferred to ICU or death within 24 hrs of identification by the EWS algorithm for intervention and control wards.
Time Frame: Within 24 hrs of an EWS alert
Measure: Number; unit: participants
Arm/Group | Control | Nurse Notification of EWS Alert
Number analyzed (Participants) | 10120 | 9911
participants | 426 | 444

2. Secondary Outcome: Clinical Outcomes and Process Measures
Description: length of stay
Time Frame: Hospital discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control | Nurse Notification of EWS Alert
Number analyzed (Participants) | 10120 | 9911
days | 6.92 [3.82 to 12.67] | 7.07 [3.99 to 12.15]

ADVERSE EVENTS:
Arm/Group | Control | Nurse Notification of EWS Alert
Serious Adverse Events (participants affected / at risk) | 0/10120 | 0/9911
Other Adverse Events (participants affected / at risk) | 0/10120 | 0/9911

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes